CLINICAL TRIAL: NCT01776944
Title: Validating a Handheld Indirect Calorimeter in Overweight and Obese Pediatric Population
Brief Title: Resting Energy Expenditure Using a Handheld Calorimeter
Acronym: CalVal
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Rajavel Elango, PhD, Principle Investigator, University of British Columbia
Other Study IDs: H12-00364
Record Dates: First submitted 2013-01-17; First posted 2013-01-28 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Obesity
Keywords: Resting energy expenditure; Handheld calorimeter; Obese and overweight; Pediatrics
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Obese children

SUMMARY:
High prevalence of obesity in children has increased associated complications such as type 2 diabetes, hypertension and fatty liver disease. Dietitians develop a meal plan that restricts caloric intake by estimating the resting and total daily energy expenditures.Estimation of energy needs is most commonly done using predictive equations. Reliable and valid energy requirements can be obtained using a traditional metabolic system, however this is an expensive option. Handheld indirect calorimeters may be a good alternative to measure energy needs. Several studies have been conducted to determine the validity and accuracy of handheld calorimeters in adults and health children, however, to the best of our knowledge, there are no such studies in the overweight and obese pediatric population.

The purpose of this study is to validate a handheld indirect calorimeter against a traditional metabolic system in overweight and obese children.

If handheld calorimeters can accurately measure resting energy expenditure in overweight and obese adolescents, dietitians will have an opportunity to tailor pediatric weight management interventions based on parameters that are unique to each individual.

ELIGIBILITY:
Inclusion Criteria:

* 13-18y of age
* BMI 85th percentile or more
* No severe illness, neurological and development issues
* not on insulin
* Able to fast overnight

Exclusion Criteria:

* not 13-18y of age
* BMI under 85th percentile
* ill or have neurological and development issues
* on insulin

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Obese children aged 13-18y of both gender
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2012-05; Primary Completion 2014-06 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Resting Energy Expenditure as measured by the traditional Indirect Calorimeter(metabolic cart) and the handheld indirect calorimeter in standardized conditions | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Rajavel Elango, Ph.D, Principal Investigator — Child & Family Research Institute/University of British Columbia
Locations (1):
- Child & Family Research Institute, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Woo P, Murthy G, Wong C, Hursh B, Chanoine JP, Elango R. Assessing resting energy expenditure in overweight and obese adolescents in a clinical setting: validity of a handheld indirect calorimeter. Pediatr Res. 2017 Jan;81(1-1):51-56. doi: 10.1038/pr.2016.182. Epub 2016 Sep 21. PMID 27653085